CLINICAL TRIAL: NCT05079503
Title: Efficacy and Safety of GEN-001 (Lactococcus Lactis) Plus Total Neoadjuvant Therapy and Dynamic Change of Gut Microbiome in Locally Advanced Rectal Cancer : Exploratory, Pilot, Prospective, Longitudinal Study
Brief Title: Gut Microbiome and Its Immune Modulation in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, SoohyeonLee, Assistant Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021AN0403
Record Dates: First submitted 2021-09-14; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNT plus GEN-001 (Experimental): Total neoadjuvant therapy (TNT) includes short-course radiotherapy (25 Gy/5fx), followed by systemic chemotherapy with FOLFOX regimen for 3-6 months. GEN-001 is orally administered once daily during total TNT periods and surgery will be performed 1 month after systemic chemotherapy.
  Interventions: Drug: GEN-001

INTERVENTIONS:
Drug: GEN-001 — GEN-001, Lactobacillus lactis is a live, purified facultative anaerobic gram-positive probiotic lactic acid bacterial strain. GEN-001 is orally administered once daily during total TNT periods.
  Other Names: Lactococcus lactis

SUMMARY:
To investigate dynamic change of gut microbiomes and metabolites, and their effects on immune modulation. To evaluate the efficacy and safety of TNT with GEN-001 (Lactococcus lactis) and identify predictive biomarkers for pathologic response in patients with locally advanced rectal cancer (LARC).

DETAILED DESCRIPTION:
The multimodality strategy, neoadjuvant chemoradiotherapy (CRT) or total neoadjuvant therapy (TNT) followed by surgery, has been widely used to improve local control and overall survival in locally advanced rectal cancer (LARC). TNT is a recently promising strategy incorporating systemic chemotherapy following short-course radiotherapy before surgery in LARC, and showed superior rates of pathologic complete response (pCR) compared with the concurrent CRT followed by surgery and adjuvant chemotherapy (CRT-A). However, issues regarding neoadjuvant therapy-related toxicity as well as disease progression during TNT have been raised, which need to identify biomarkers for prediction of treatment responses and safety in patients with LARC.

Growing evidence suggests that gut microbiomes interact with tumor microenvironment and are related with inflammation and immunomodulation. The association between gut microbiomes and responses of chemotherapy or immunotherapy has been previously reported. The administration of certain beneficial microbiome can be one of the strategies to treat gut dysbiosis in cancer patients, restoring microbial diversity and changing the composition of microbiome. GEN-001, Lactobacillus lactis is a live, purified facultative anaerobic gram-positive probiotic lactic acid bacterial strain. The preclinical studies showed the potential therapeutic effects of GEN-001 as an anti-cancer treatment through the activation of immune cells, including CD4 or CD8 T-cells and natural killer cells, and synergistic effects with oxaliplatin chemotherapy. Therefore, the investigators plan to investigate dynamics of gut microbiomes and metabolites, and their effects on immune modulation. Additionally investigators plan to evaluate the efficacy and safety of TNT with GEN-001 and identify predictive biomarkers for pathologic response in patients with LARC.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 19 years
2. Locally advanced rectal cancer, histologically confirmed; clinically T3/4, clinically N+, enlarged lateral lymph nodes, extramural vascular invasion (+), or mesorectal fascia (+)
3. Patients who schedule to receive total neoadjuvant therapy, including short-course radiotherapy (25 Gy in 5 fractions), followed by FOLFOX chemotherapy (5-fluorouracil, leucovorin, and oxaliplatin)
4. Patients with ability to swallow and retain oral medication and no clinically significant gastrointestinal abnormalities that may alter absorprtion
5. Patients with ability to collect their blood and stool samples

Exclusion Criteria:

1. Rectal cancer, other histologic type than adenocarcinoma (such as squamous cell carcinoma)
2. Patients who schedule to receive concurrent chemoradiotherapy or short-course radiotherapy alone followed by surgery and adjuvant chemotherapy
3. Patients who need emergent surgery or colostomy due to obstruction or bleeding
4. Prior use of proton pump inhibitors or H2 blockers, probiotics, immunosuppressive agents, and antibiotics within 4 weeks
5. Patients have concurrent medication that may interact with fluoropyrimidine or oxaliplatin (i.e. flucytosine, phenytoin, or warfarin)
6. Known prior history of severe adverse events during fluoropyrimidine or deficiency of dihydropyrimidine dehydrogenase (DPD)
7. Known prior severe hypersensitivity to platinum
8. Patients who have an active infection requiring antibiotics, antifungal, or antiviral agents
9. Prior solid organ or allogenic stem cell transplantation

11. Patients who have clinically significant medical disease

* Cardiovascular disease <6 months prior to enrollment (myocardial infarction, unstable angina, coronary artery bypass surgery or percutaneous coronary intervention)
* Cerebral vascular accident/stroke (<6 months prior to enrollment)
* Congestive heart failure (≥New York Heart Association (NYHA) Classification Class II)
* Uncontrolled hypertension by standard therapy: systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg
* Serious cardiac arrhythmia requiring medication 12. Pregnant women 13. Patients who have psychiatric condition that would prohibit the understanding or rendering of informed consent or that would limit compliance with study requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic change of gut microbiome: a-diversity index | up to 30 weeks
  16s rRNA sequencing
Dynamic change of gut microbiome: b-diversity index | up to 30 weeks
  16s rRNA sequencing
Immune modulation in blood | up to 30 weeks
  Cytotoxic T cells or regulatory T cells using flowcytometry
Immune modulation in tissue | up to 30 weeks
  CD4 or CD8 tumor-infiltrating lymphocytes using immunohistochemistry

SECONDARY OUTCOMES:
Efficacy and safety of TNT plus GEN-001 | up to 30 weeks
  Achieving pathologic complete response
Identify predictive biomarkers for pathologic responders | up to 30 weeks
  Prediction for pathologic complete response

IPD SHARING:
Plan to Share IPD: No